CLINICAL TRIAL: NCT05391607
Title: Randomized Trial of Intraoperative Intravascular Effect of Hyper-oncotic 20% Albumin, Iso-oncotic 5% Albumin and Ringer Lactate During Haemorrhage in Cystectomy. A Prospective Randomized Active-controlled Single Centre Trial
Brief Title: Comparison Between Hyperoncotic and Isooncotic Albumin to Support Blood Loss Replacement
Acronym: VASCALB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VASCALB
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-05

CONDITIONS: Blood Loss, Surgical; Fluid Retention
Keywords: hyperoncotic; isooncotic; albumin 20%; albumin 5%; ringer lactate; blood loss; hemorrhage; fluid replacement; intravascular effect; volume expansion; cystectomy; pro-ANP; pro-BNP; glycocalyx proteins; microcirculation damages; endothelial shedding; CD138/syndecan 1; heparan sulfate; hyaluronic acid
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage | interventions — galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20; zidovudine 5'-monophosphate-mannose-albumin conjugate; Control Groups; Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Albumin 20% (Experimental): 3mL/kg (ideal body weight) completed by a Ringer-lactate crystalloid ratio 1:1 to total amount of blood loss during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Interventions: Drug: Hyperoncotic Albumin 20%
- Albumin 5% (Experimental): 12ml/kg (ideal body weight) completed by a Ringer-lactate crystalloid ratio 1:1 to total amount of blood loss during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Interventions: Drug: Isooncotic Albumin 5%
- Ringer-lactate (Active Comparator): Ratio 3:1 of total of blood loss during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Interventions: Drug: Ringer's Lactate Crystalloid Solutions (control group)

INTERVENTIONS:
Drug: Hyperoncotic Albumin 20% — Intravenous administration during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Other Names: Albumin 20%
  Arms: Albumin 20%
Drug: Isooncotic Albumin 5% — Intravenous administration of Albumin 5% 12ml/kg (ideal body weight) completed by a Ringer-lactate crystalloid ratio 1:1 to total amount of blood loss during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Other Names: Albumin 5%
  Arms: Albumin 5%
Drug: Ringer's Lactate Crystalloid Solutions (control group) — Intravenous administration of Ringer-lactate ratio 3:1 of total of blood loss during removal of the bladder (i.e. the bleeding part) of cystectomy procedures.
  Other Names: Ringer Lactate
  Arms: Ringer-lactate

SUMMARY:
Fluid intravascular replacement is usually performed with either balanced crystalloids or iso-oncotic colloids, (synthetic colloids, plasma and 5% albumin). Doubts have been raised about synthetic colloids, and albumin solutions have been used more extensively. Albumin is the main protein responsible for plasma oncotic pressure and its volume expansion effect. The mobilization of extravascular fluid by infusing a hyper-oncotic solution like 20% albumin solution has been shown, causing endogenous fluid recruitment and blood volume expansion.

The primary objective of this study is to compare the effect on plasma volume expansion and fluid recruitment of 3 different types of fluids (Albumin 5% and Albumin 20% and Ringer-lactate) during the hemorrhagic phase of the cystectomy procedure.

Secondary objectives are the assessment of the hemodynamic parameters during surgery and the follow-up of pro-ANP and pro-BNP peptides. Glycocalyx proteins will be followed to evaluate endothelial wall shedding and microcirculation damages.

DETAILED DESCRIPTION:
Bladder cancer occurs mainly in old comorbid patients. The standard treatment of localized muscle invasive bladder cancer is pelvic lymph node dissection and radical cystectomy with urinary diversion. Optimal perioperative fluid management for this surgery is challenging and still controversial in terms of how much to perfuse, choice of fluids to restore hydrated state and volemia.

Fluid treatment is usually performed with either balanced crystalloids fluids or iso-oncotic synthetic colloids, or albumin 5%. Because crystalloids quickly equilibrate between the intravascular and interstitial volumes, they are mainly used to treat dehydration and temporary volume deficits. Doubts have been raised about synthetic colloids and the natural albumin has been used more extensively. Albumin is the main protein responsible for plasma oncotic pressure and its volume expansion effect.

Iso-oncotic colloids (Albumine 5%) remain intravascular for a prolonged period, but they play a neutral role in terms of endogenous fluid recruitment, as the oncotic pressure is equilibrated between the intra- and extra- vascular territories.

An alternative therapeutic option is the mobilization of tissue fluid by infusing a small amount of hyper-oncotic fluid like the albumin 20% solution, which has showed the advantage in its blood volume expansion capacities over crystalloids (endogenous fluid recruitment).

The effects of the Albumin 20% solution have until now never been compared in a same perioperative setting to the Albumin 5% nor to Ringer-lactate solution.

The investigators will evaluate the physiological effects and their outcomes between these fluid therapies in the frame of blood loss replacement during the hemorrhagic part of cystectomy procedures. The investigators will as well assess the variation of hemodynamic parameters (pro-ANP, pro-BNP) and the resulting microcirculation damages (endothelial wall shedding).

ELIGIBILITY:
Inclusion Criteria:

* Non emergent radical cystectomy with urinary diversion
* Adult: older than 18 years
* Written informed consent

Exclusion Criteria:

* Contraindications to the class of drugs under study (i.e: known hypersensitivity/ allergy to class of drugs or to the investigational product).
* Renal insufficiency: GFR: <60ml/min/1.73m2 (KDIGO Clinical Practice Guideline for Acute Kidney Injury, stage 3 and over).
* History of heart failure.
* Use of diuretic treatment.
* Women who are pregnant or breast feeding (exclusion of surgery per se).
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Plasma volume expansion | 5 hours
  Difference in plasma volume expansion of albumin 20%, albumin 5% and Ringer lactate calculated by volume kinetics

SECONDARY OUTCOMES:
Biological markers (pro-ANP and pro-BNP) | 24 hours
  Variation and comparison of kinetics hemodynamics biological markers such as pro-ANP and pro-BNP
Cardiac output (CO) | 5 hours
  Evolution of cardiac output (CO) at the start of surgery, begin of infusion, stop of infusion and end of surgery.
Endothelial damage | 24 hours
  Assessment of microcirculation damage due to peroperative stress and fluid therapy through Glycocalyx proteins (CD-138/syndecan 1, heparan sulfate and hyaluronic acid).
Stroke volume (SV) | 5 hours
  Evolution of stroke volume at the start of surgery, begin of infusion, stop of infusion and end of surgery.
Pleth variability index (PVI) | 5 hours
  Evolution of pleth variability index (PVI) at the start of surgery, begin of infusion, stop of infusion and end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wuethrich, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Patrick Wuethrich, Department of Anaesthesiology and Pain Therapy, University Hospital Bern Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jardot F, Hahn RG, Huber M, Wuethrich PY. Detection of hypovolemia by non-invasive hemodynamic monitoring during major surgery using Ringer s solution, 5% albumin, or 20% albumin as infusion fluid: a post-hoc analysis of a randomized clinical trial. Crit Care. 2025 Mar 23;29(1):132. doi: 10.1186/s13054-025-05357-z. PMID 40122881
- [Derived] Jardot F, Hahn RG, Engel D, Beilstein CM, Wuethrich PY. Blood volume and hemodynamics during treatment of major hemorrhage with Ringer solution, 5% albumin, and 20% albumin: a single-center randomized controlled trial. Crit Care. 2024 Feb 5;28(1):39. doi: 10.1186/s13054-024-04821-6. PMID 38317178